CLINICAL TRIAL: NCT00653393
Title: To Compare Bioavailability of Kali Tranylcypromine 10mg Tablets to That of Parnate 10 mg Tablets Under Fasting Conditions.
Brief Title: Bioavailability Study of Tranylcypromine 10mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: SFBC Ft. Myers, Inc (Industry)
Responsible Party: Dr. Alfred Elvin/ Director Biopharmaceutics, Par Pharmaceutical, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 04-0413-001
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2008-04

CONDITIONS: To Determine the Bioavailability of Tranylcypromine
Keywords: bioequivalence, single- dose, fasting
MeSH Terms: conditions — Fasting | interventions — Tranylcypromine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects received Kali product under fasting conditions
  Interventions: Drug: Tranylcypromine
- B (Active Comparator): Subjects received Parnate product under fasting conditions
  Interventions: Drug: Parnate

INTERVENTIONS:
Drug: Tranylcypromine — Tablets, 10 mg, single-dose
  Other Names: Parnate
  Arms: A
Drug: Parnate — Tablets, 10 mg, single-dose
  Other Names: Tranylcypromine
  Arms: B

SUMMARY:
To compare the single-dose Bioavailability of Tranylcypromine and Parnate

DETAILED DESCRIPTION:
To compare the relative Bioavailability of Tranylcypromine 10 mg tablets with that of PARNATE 10mg tablets in normal,healthy, men and women under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be normal, healthy adult men and women who volunteer to participate.
* Is the individual healthy, nonsmoking, normal adult man or woman who volunteers to participate?
* Is s/he at least 18 years of age? Is his/her BMI between 19 and 30, exclusive?
* Is she willing to avoid pregnancy by abstaining from sexual intercourse, or by the use of barrier methods. (diaphragm, condom, foams/jellies, sponge), and IUD, or has she has been surgically sterile or post- menopausal at least six months prior to entering into the study?
* Is s/he considered reliable and capable of understanding his/her responsibility and role in the study?
* Has/s/he provided written informed consent?
* A no answer to any of the above questions indicates taht the individual is ineligible for enrollment.

Exclusion Criteria:

* Does the individual have a history of allergy or hypersensitivity to tranylcypromine?
* Does/ s/he have clinically significant laboratory abnormalities that would interface with the conduct or interpretation of the study or jeopardize his/her safety?
* Does s/he have significant history or clinical evidence of auto-immune, cardiovascular, gastrointestinal, hematopoietic, hepatic, neurological, ongoing infection, pancreatic, or renal diseases that would interface with the conduct or interpretation of the study or jeopardize his/her safety?
* Is she nursing?
* Does s/he have serious psychological illness?
* Does s/he have significant history ( within the past year) or clinical evidence of alcohol or drug abuse?
* Does s/he have a positive urine drug screen or saliva alcohol screen, or a positive HIV-1 , or hepatitis B or C screen, or a positive pregnancy test?-Is s/he unable to refrain from the use of alcohol or xanthine-containing foods or beverages during periods beginning 48 hours prior to study drug administration and ending when the alst blood sample has been taken?
* Is s/he unable to refrain from the ingestion of smoked meat, cheese (except cream cheese and cottage cheese), wine and beer during periods beginning 48 hours prior to study initiation and ending seven days after the last blood sample has been taken in study period two?
* Has s/he used any prescription drug during the 14-day period prior to study initiation, or any OTC drug during the 72-hour period preceding study initiation?
* Is s/he unable to refrain from the use of all concomitant medications during the study?
* Ha s/he donated or lost blood, or participated in a clinical study which involved the with drawl of a large volume of blood (480mL or more), during the six week period preceding study initiation?
* Has s/he donated an investigational drug during the 30 day period preceding study initiation?
* A yes answer to any of the above questions indicates that the individual is ineligible for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-10; Primary Completion 2004-11 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pizzaro, Principal Investigator — SFBC Ft. Myers, Inc
Locations (1):
- SFBC Ft. Myers, Inc, Fort Myers, Florida, United States